CLINICAL TRIAL: NCT06517914
Title: A First-in-Human, Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Following Oral Administration of YH35995 in Healthy Adult Male Participants
Brief Title: A First-in-Human, Single- and Multiple-Ascending Dose Study of YH35995 in Healthy Adult Male Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YH35995-101
Record Dates: First submitted 2024-07-14; First posted 2024-07-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: YH35995; Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study, meaning that YH35995 tablets and placebo tablets will be identical in appearance and will be packaged in the same way.
  Information about the treatment arm to which participants are assigned must remain blinded for the duration of the study unless information about the causal relationship between the adverse event and the Investigational Product that meets the drug withdrawal criteria becomes essential or, in an emergency, if the information about the Investigational Product becomes critical for treating the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YH35995 (Experimental): [Part A] Participants will be orally administered a single dose of YH35995 in five dose groups, gradually escalating from lower to higher doses. Each cohort includes 10 participants (8 randomly assigned to the YH35995 arm and 2 randomly assigned to the placebo arm).
  [Part B] Participants will receive multiple oral doses of YH35995 once every 4 weeks in three dose groups. Each cohort includes 12 participants (9 randomly assigned to the YH35995 arm and 3 randomly assigned to the placebo arm).
  Interventions: Drug: YH35995
- Placebo (Placebo Comparator): [Part A] Participants will be orally administered a single dose of Placebo in five dose groups, gradually escalating from lower to higher doses. Each cohort includes 10 participants (8 randomly assigned to the YH35995 arm and 2 randomly assigned to the placebo arm).
  [Part B] Participants will receive multiple oral doses of Placebo once every 4 weeks in three dose groups. Each cohort includes 12 participants (9 randomly assigned to the YH35995 arm and 3 randomly assigned to the placebo arm).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YH35995 — Oral administration of YH35995
  Arms: YH35995
Drug: Placebo — Oral administration of Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, first-in-human study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of single and multiple oral doses of YH35995

DETAILED DESCRIPTION:
YH35995 is being developed as a treatment for the neurological symptoms of Gaucher Disease type 3. This study is a first-in-human (FIH), phase 1, randomized, double-blind, placebo-controlled study of YH35995, which consists of two parts. In Part A (SAD), single ascending dose of YH35995 is administered to healthy male participants to assess its safety, tolerability, PK, and PD. In Part B (MAD), multiple ascending dose of YH35995 is administered to healthy male participants to assess its safety, tolerability, PK, and PD.

ELIGIBILITY:
Inclusion Criteria:

* Male between the ages of 19 and 45 at the time of providing written consent
* Participants who weigh at least 50 kg at screening and have a body mass index (BMI) of at least 18.0 kg/m2 and less than 30 kg/m2
* Participants who have been fully informed about and fully understand this study, have voluntarily decided to participate, and have agreed in writing to comply with the guidelines of the study during the duration of the study

Exclusion Criteria:

* Participation in a bioequivalence trial or any other clinical trials within 6 months prior to the first scheduled dose of the IP (within 1 month of the first scheduled dose for participants who have taken part in a dietary supplement clinical trial)
* Individuals with clinically significant abnormal results that do not match any other inclusion/exclusion criteria, as determined by the principal investigator and the delegated persons(investigator)
* Individuals who are unwilling or unable to comply with the participant guidelines described in this protocol

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
[Part A, B] Treatment-emergent adverse events (TEAEs) | Part A: Day1-150, Part B: Day1-232
  To assess the safety and tolerability of a single dose and multiple dose administration of YH35995

SECONDARY OUTCOMES:
[Part A] Maximum observed plasma concentration (Cmax) | Day1-150
  To characterize the pharmacokinetics (PK) of YH35995
[Part A] Time to reach Cmax (Tmax) | Day1-150
  To characterize the pharmacokinetics (PK) of YH35995
[Part A] Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | Day1-150
  To characterize the pharmacokinetics (PK) of YH35995
[Part A] AUC from time 0 to infinity (AUCinf) | Day1-150
  To characterize the pharmacokinetics (PK) of YH35995
[Part A] Apparent terminal elimination half-life (t1/2) | Day1-150
  To characterize the pharmacokinetics (PK) of YH35995
[Part A] Total plasma clearance (CL/F) | Day1-150
  To characterize the pharmacokinetics (PK) of YH35995
[Part A] Apparent volume of distribution (Vz/F) | Day1-150
  To characterize the pharmacokinetics (PK) of YH35995
[Part B] Cmax during the first dosing interval | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Tmax during the first dosing interval | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] AUC during the first dosing interval (AUCsingle) | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] AUC during the dosing interval at steady state (AUCtau,ss) | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Cmax at steady state (Cmax,ss) | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Tmax at steady state (Tmax,ss) | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Accumulation ratio using AUC (Rac(AUC)) | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Accumulation ratio using Cmax (Rac(Cmax)) | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Plasma concentration at the last observed time point during the dosing interval at steady state (Ctrough) | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Average plasma concentration (Cavg) | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Clearance at steady state (CLss/F) | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Volume of distribution at steady state (Vss) | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Effective half-life (t1/2,Rac) | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Cerebrospinal fluid to plasma concentration ratio(C/P ratio) of YH35995 | Day1-232
  To assess the pharmacokinetics (PK) of YH35995 after multiple dose administration
[Part B] Properly derived PD parameters for YH35995, including the area under the effect curve (AUEC) and maximum effect (Emax) | Day1-232
  To assess the pharmacodynamics (PD) of YH35995 after multiple dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Hyounggyoon Yoo, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA Bundang Medical Center, Seongnam, Bundang-gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including data dictionaries) that underline the results reported in study-related publications will be made available during the period beginning 1 year and ending 5 years after all trial primary and secondary endpoints were assessed. Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to clinicaltrials@yuhan.co.kr.
  A summary of the study results will be posted in the publicly accessible database (i.e. clinicaltrials.gov) no later than 1 year after the study's primary completion date.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 1 year and ending 5 years after all trial endpoints were assessed
Access Criteria: Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to clinicaltrials@yuhan.co.kr